CLINICAL TRIAL: NCT01735747
Title: Phase Ⅱ Trial of Temozolomide Plus Concurrent Whole-Brain Radiation Followed by TNV Regimen as Adjuvant Therapy for Patients With Newly Diagnosed Primary Central Nervous System (CNS) Lymphoma (PCNSL)
Brief Title: Temozolomide, Nedaplatin, Vincristine, and Radiotherapy as First-line Treatment in Newly Diagnosed Primary CNS Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rongjie Tao (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Rongjie Tao, Neurosurgery, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI 002
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Central Nervous System Tumors
Keywords: Lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma | interventions — Radiotherapy; Chemoradiotherapy; nedaplatin; Vincristine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide, Nedaplatin, Vincristine, Radiotherapy (Experimental): The newly diagnosed PCNSL patients will be given concurrent temozolomide (75mg/m2, orally) daily during WBRT. Then, the TNV regimen will be given after four weeks. TNV regimen consisted of temozolomide (200mg/m2 orally, days 1-5), nedaplatin (80mg/m2 i.v., day 1), vincristine (1.4mg/m2 i.v., day 1). Each cycle was 4 weeks and a maximum of six cycles were applied.
  Interventions: Radiation: Radiotherapy; Drug: nedaplatin; Drug: vincristine; Drug: Temozolomide

INTERVENTIONS:
Radiation: Radiotherapy — WBRT was given five times a week at 2 gray (Gy)/d until the whole brain radiotherapy dose reached 40 gray. The patients were given concurrent temozolomide (75mg/m2, orally) daily during radiotherapy until the end of radiotherapy.
  Other Names: WBRT (whole-brain radiotherapy); Concurrent Chemoradiotherapy
Drug: nedaplatin — nedaplatin (80mg/m2 i.v., day 1), 28 day schedule, performed four weeks after radiotherapy.A maximum of six cycles were applied.
Drug: vincristine — vincristine (1.4mg/m2 i.v., day 1)28 day schedule,performed four weeks after radiotherapy.A maximum of six cycles were applied.
  Other Names: ao-xian-da
Drug: Temozolomide — Temozolomide (200mg/m2 orally, days 1-5, Each cycle was 4 weeks ), performed four weeks after radiotherapy. A maximum of six cycles were applied.

SUMMARY:
In this trial, we will treat newly diagnosed PCNSL with temozolomide, nedaplatin, vincristine (TNV) as the replacement of high-dose methotrexate to combine with concurrent chemoradiotherapy. Our objective was to assess our treatment strategies' availability based on response rates, progression-free survival (PFS), median PFS, and toxicity.

DETAILED DESCRIPTION:
The best reported outcomes of PCNSL treatment are high-dose methotrexate-based chemotherapy combined with whole-brain radiation therapy (WBRT). Despite aggressive therapy, however, nearly 50% of patients will relapse within 24 months of diagnosis. Furthermore, the application of high-dose methotrexate-based regimen is complex, needing be hydrated, alkalified and detoxified, and treatment-related toxicity mortality is severe[3,4]. In an attempt to improve upon these poor results and reduce treatment-related side effects, we will treat about 15-20 PCNSL patients with temozolomide concurrent chemoradiotherapy at the outset and then adjuvant chemotherapy for 6 cycles with temozolomide, nedaplatin, vincristine, as part of front-line therapy. Our objective is to assess our treatment strategies' availability based on response rates, progression-free survival (PFS), median PFS, and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary CNS lymphoma.
* Newly diagnosed.
* ECOG (Eastern Cooperative Oncology Group) Performance status of 0-1.
* Relevant hospital examination including laboratory examination and physical examination (Chest X-ray, electrocardiogram, abdomen B ultrasonography, magnetic resonance imaging (MRI) of head and neck) must to be done, in order to exclude other system fatal diseases.
* Must have adequate organ function as defined by the protocol: Adequate renal function: serum creatinine ≤ 1.5 mg/dl and/or calculated creatinine clearance ≥ 60 ml/min; Adequate hepatic function: bilirubin level ≤ 1.5 x ULN, ASAT & ALST ≤ 1.5 x ULN.Adequate bone marrow reserves: neutrophil (ANC) count ≥ 1500 /mm^3, platelet count ≥ 100,000 /mm^3, hemoglobin ≥ 9 g/dl.
* Age >/= 18 and </= 75 years
* Signed written informed consent prior to study entry.

Exclusion Criteria:

* Patients with human immunodeficiency virus seropositivity and systemic lymphoma manifestation.
* Serious uncontrolled concurrent illness.
* Previous brain radiotherapy, systemic chemotherapy.
* Concurrent chronic systemic immune therapy, targeted therapy not indicated in this study protocol.
* Any evidence of prior exposure to Hepatitis B virus.
* Unable to comprehend the study requirements or who are not likely to comply with the study parameters.
* Pregnant (confirmed by serum or urine β-HCG) or lactating.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-06; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Rate of complete radiologic response (CR) | 3 years
  final data collection date for primary outcome measure

SECONDARY OUTCOMES:
Failure-free survival | 3 years
Toxicity | 3 years
Overall response rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yu-fang Zhu, M.D., Study Director — Shandong Cancer Hospital and Institute; Yong Wang, M.M., Study Director — Shandong Cancer Hospital and Institute
Locations (1):
- Neurosurgery, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

REFERENCES:
- [Background] Reni M, Zaja F, Mason W, Perry J, Mazza E, Spina M, Bordonaro R, Ilariucci F, Faedi M, Corazzelli G, Manno P, Franceschi E, Pace A, Candela M, Abbadessa A, Stelitano C, Latte G, Ferreri AJ. Temozolomide as salvage treatment in primary brain lymphomas. Br J Cancer. 2007 Mar 26;96(6):864-7. doi: 10.1038/sj.bjc.6603660. Epub 2007 Feb 27. PMID 17325700
- [Background] Kurzwelly D, Glas M, Roth P, Weimann E, Lohner H, Waha A, Schabet M, Reifenberger G, Weller M, Herrlinger U. Primary CNS lymphoma in the elderly: temozolomide therapy and MGMT status. J Neurooncol. 2010 May;97(3):389-92. doi: 10.1007/s11060-009-0032-0. Epub 2009 Oct 20. PMID 19841864
- [Background] DeAngelis LM, Seiferheld W, Schold SC, Fisher B, Schultz CJ; Radiation Therapy Oncology Group Study 93-10. Combination chemotherapy and radiotherapy for primary central nervous system lymphoma: Radiation Therapy Oncology Group Study 93-10. J Clin Oncol. 2002 Dec 15;20(24):4643-8. doi: 10.1200/JCO.2002.11.013. PMID 12488408